CLINICAL TRIAL: NCT04649281
Title: Insomnia and Sleep Disturbances in Chronic Pain Patients - Relation to Physical Activity Level and Opioid Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 272924
Record Dates: First submitted 2020-10-28; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain; Insomnia; Exercise; Sleep; Sleep Disorder; Opioid Use
Keywords: Accelerometry; Mental fatigue; Self-Efficacy
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders; Motor Activity; Sleep Wake Disorders; Mental Fatigue | interventions — Accelerometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerometry (Other): Recording of sleep and physical activity by accelerometry during one week.
  Interventions: Device: Accelerometry

INTERVENTIONS:
Device: Accelerometry — Recording of sleep and physical activity by accelerometry during one week.

SUMMARY:
Pain is one of the most common causes of healthcare contact and long-term sick leave, with negative consequences on physical and mental health. Poor sleep is common in chronic pain patients. Epidemiological studies indicate that 5-7% of patients with chronic pain are treated regularly with strong opioids. Negative side effects of pain modulating drugs on sleep quality have been reported, which may have negative influence on overall disease management in chronic pain patients. However, to date there are conflicting results regarding the effects of opioids on sleep, since the pain relieving effect of opioids seem to affect sleep positively. There is data suggesting that physical activity has positive effects on both pain perception and sleep quality (and duration). The aim of the study is to explore insomnia and characteristics of sleep in patients with chronic pain and the relationship with physical activity level and opioid use.

DETAILED DESCRIPTION:
One hundred participants with planned follow-up (decision according to clinical routine) at the Pain Centre will be consecutively recruited. After signed informed consent, the participants will wear two accelerometers during one week, one for recording sleep and one for recording physical activity. The participants will be asked to fill out a sleep and pain diary during the same week. Furthermore, the participants will fill out questionnaires regarding sleep, life style, mental fatigue and self-efficacy. All study participant are included in the Swedish Quality Registry for Pain Rehabilitation (SQRP). Data from the SQRP will be used regarding patient health characteristics, pain and pain associated symptoms, health related quality of life, sleep and self-reported physical activity level. Data regarding co-morbidity, drug use, pharmacological treatment and other interventions at the Pain Center will be collected from the patient charts. In addition, the participants blood pressure and neck circumference will be measured. Blood samples will be analysed for biomarkers associated with pain and sleep disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain (i.e. pain > 3 months)
* Planned follow up at the Pain Centre
* Age ≥18 years
* Consents to participation in the study

Exclusion Criteria:

* Inadequate knowledge of the Swedish language
* Alcohol or substance abuse
* Severe untreated psychiatric disorders including psychiatric disease and/or psychological conditions which are the primary determinant to the patient's pain condition
* Malignant disease with short expected survival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep | Daily assessment during one week
  Sleep duration in minutes assessed by accelerometry
Sleep | Daily assessment during one week
  Sleep timing, i.e. sleep onset and wake time assessed by accelerometry
Physical activity | Daily assessment during one week
  Minutes of physical activity per week at moderate and vigorous intensity physical activity (MVPA), minutes of sedentary behaviour (SED) assessed by accelerometry
Opioid consumption | Opioid consumption at study enrollment
  Opioid consumption in morphine equivalent doses
Pain intensity | Daily assessment during one week
  Pain intensity according to Numeric Rating Scale (NRS), score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable"

SECONDARY OUTCOMES:
Insomnia Severity | Insomnia severity at enrollment
  Total Score from the 7-item Insomnia Severity Index where total score ranges from 0-28 and higher scores indicate greater severity of insomnia.
Sleep quality | Sleep quality at study enrollment
  Assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 self-rated questions which assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep related problems. The 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The seven component score are then summed to yield a global PSQI score which has a range of 0-21; higher scores indicate worse sleep quality.
Daytime sleepiness | Daytime sleepiness at study enrollment
  Epworth Sleepiness Scale (ESS), which quantifies daytime sleepiness. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher daytime sleepiness.
Self-assessed physical activity | Self-assessed physical activity at study enrollment
  Minutes of physical activity per week (physical exercise and daily exercise) and minutes of sedentary behaviour per week.
Self-efficacy for exercise scale | Self-efficacy for exercise at study enrollment
  The Self-efficacy for exercise scale measures a patient's self-efficacy when it comes to physical exercise. The questionnaire consists of 9 questions that can be answered on a 1-10 scale. A total score between 9 and 90 is calculated, were a higher number represent a better outcome.
Mental fatigue scale | Mental fatigue at study enrollment
  The mental fatigue scale (MFS) is a multidimensional questionnaire containing 15 questions. A total score between 0-42 is calculated. A score >10 indicates a problem with mental fatigue.
Sleep dairy | Daily assessment during one week
  Self-assessed sleep latency, total sleep time, wake time after sleep onset and sleep quality.

OTHER OUTCOMES:
Neurofilament light | Neurofilament light at study enrollment
  Neurofilament light in blood sample
25-hydroxyvitamin D | 25-hydroxyvitamin D at study enrollment
  Levels of Serum 25-hydroxyvitamin D (25[OH]D)

CONTACTS AND LOCATIONS:
Overall Officials: Paulin Andréll, MD, PhD, Principal Investigator — Sahlgrenska University Hospital, Region Västra Götaland; Göteborg University
Locations (1):
- Pain Centre, Department of Anaesthesiology and Intensive Care Medicine Östra, Sahlgrenska University Hospital, Region Västra Götaland, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No